CLINICAL TRIAL: NCT06395493
Title: A 12-week Pilates Programme for Low Back Pain: Perceived and Actual Outcomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malta (Other)
Responsible Party: Principal Investigator, Janette Falzon, Principal Investigator, University of Malta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FHS-2023-00546
Record Dates: First submitted 2024-04-24; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Low Back Pain
Keywords: Pilates; Exercise; Low Back Pain; Duration; Quality of Life; Disability; Anxiety
MeSH Terms: conditions — Low Back Pain; Motor Activity; Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pilates Intervention Group (Experimental): The Pilates intervention group will consist of a twice weekly sessions for a duration of 1 hour each for a period of 12 weeks. These sessions will be conducted at the Physiotherapy Department at St Luke's Hospital and the physiotherapist, who is the main researcher will be leading the Pilates sessions.
  Interventions: Procedure: Pilates Group
- Exercise Intervention Group (Experimental): The exercise group will also receive a twice weekly session, each lasting 1 hour for a duration of 12 weeks. This group will be assigned general exercises for the low back, which will also be supervised and directed by the primary researcher.
  Interventions: Procedure: Exercise Group
- Control Group (Experimental): The control group, on the other hand will include patients who either opt not to do the exercises or are on the waiting list for physiotherapy treatment. However, after completing the 12 weeks of no intervention, they will be asked whether they would like to receive physiotherapy treatment.
  Interventions: Procedure: Control Group

INTERVENTIONS:
Procedure: Pilates Group — In this study, the participants in the Pilates group will undergo 2 sessions per week, for 12 consecutive weeks.
  Arms: Pilates Intervention Group
Procedure: Exercise Group — In this study, the participants in the Exercise group will undergo 2 sessions per week, for 12 consecutive weeks.
  Arms: Exercise Intervention Group
Procedure: Control Group — The participants in the control group, are those who either opt not to do the exercises or are on the waiting list for physiotherapy intervention. Therefore, they will not undergo any intervention for 12 consecutive weeks.
  Arms: Control Group

SUMMARY:
Pilates has emerged as a prominent exercise therapy gaining recognition among healthcare professionals for its potential benefits in managing low back pain (LBP). As healthcare practitioners increasingly incorporate Pilates into clinical practice, understanding its effects on LBP becomes crucial. This study explores the rationale behind Pilates as a therapeutic intervention for LBP, its diverse applications, varying programme durations, and the significance of long-term follow-ups. Through an examination of existing studies, the aim is to unravel the nuanced impact of Pilates on pain intensity, functional disability, and overall quality of life for individuals experiencing LBP. Furthermore, this study addresses gaps in current research, guiding the way for an extended exploration into the ideal duration of Pilates programmes and the implications of sustained, long-term engagement.

Throughout this research study, the following research question was adopted: What is the perception and actual outcomes of a Pilates programme in the management of LBP in the short and long term?

The null hypothesis (H0) for this study was that there is no significant difference following a 12 weeks Pilates programme in all outcome measures. The alternative hypothesis (H1) stated that there is significant difference in outcomes following a 12-week Pilates programme in the management of LBP.

DETAILED DESCRIPTION:
The study will investigate a longitudinal, observational three armed, interventions about the effectiveness of the 12-week pilates programme. The study will be divided in 2 phases. The first phase will seek the perception of people on Pilates in the treatment of LBP using the self-designed Questionnaire 1. The first part of the questionnaire will inquire about their experience with LBP, while the second part will involve questions regarding Pilates as a therapeutic approach.

For the first phase of the study, a minimum number of 140 participants will take part in the study. This was calculated on a total sample of 1052 patients referred for physiotherapy treatment with LBP in the year 2022. A physiotherapist from the Physiotherapy Department at the rehabilitation hospital in-charge of the back clinic shall act as an intermediary. The intermediary will contact the participants in order to deliver Questionnaire 1 either via email or postal mail before the start of any physiotherapy intervention. The questionnaires will be returned to the intermediary based on how they were originally sent, either via email or postal mail, according to the participant's choice. These questionnaire will then be passed on to the researcher for analysis. To ensure participant anonymity, the questionnaires will be coded. The intermediary will be responsible for securely managing and retaining the assigned codes.

The second phase of the study will be the intervention part. A total of 90 participants, who have completed the first phase of the study, will be randomly assigned by an intermediary, who is a physiotherapist, in change of the back clinic at the Physiotherapy Department at St Lukes' Hospital, by using a computer random generator. Simple randomization will be carried out to randomly allow each participant to either one of the 3 groups, that is the Pilates, Exercise or Control group using a computer random generator. This will ensure equal probability of assigning the participants to any group.

Prior to the Pilates intervention, all participants will be screened by the following 4 outcome measures: Numeric Pain Rating Scale (NPRS), Quebec Back Pain Disability Scale (QBPDS), RAND 36-Item Health Survey and Hospital Anxiety and Depression Scale (HADS). All outcome measures will be assessed at baseline, 4-weeks, 8-weeks, 12-weeks and then again at 24 weeks and 52-weeks post the intervention. To mitigate participant attrition rates, particularly after completing the 12-weeks programme when clinic attendance may become challenging, all outcome measures will be conducted via telephone interviews.

In the second phase of the study, the Pilates intervention group will consist of a twice weekly sessions for a duration of 1 hour each for a period of 12 weeks. These sessions will be conducted at the Physiotherapy Department at St Luke's Hospital and the physiotherapist, who is the main researcher will be leading the Pilates sessions. The exercise group will also receive a twice weekly session, each lasting 1 hour for a duration of 12 weeks. This group will be assigned general exercises for the low back, which will also be supervised and directed by the primary researcher. The control group, on the other hand will include patients who either opt not to do the exercises or are on the waiting list for physiotherapy treatment. However, after completing the 12 weeks of no intervention, they will be asked whether they would like to receive physiotherapy treatment.

After completing the Pilates intervention group, participants will be given Questionnaire 2 to review the perception of Pilates following the intervention. This questionnaire will specifically address Pilates as a treatment method. By comparing the responses from Questionnaire 1 with the feedback obtained from Questionnaire 2, this study aim to assess the alignment between participants' perceptions of Pilates and their actual experiences following the intervention. The questionnaires will be distributed and collected by hand by the intermediary on the last day of intervention.

Both questionnaires will be coded in order to ensure the participants' anonymity and the intermediary will be responsible for securely managing and retaining the assigned codes.

ELIGIBILITY:
Inclusion Criteria:

* Participants between the age of 18-65
* Participants who have been experiencing LBP for more than 3 months
* Participants who have not undergone surgical intervention for their back in the past 6 months
* Participants who were willing to attend the Pilates programme twice a week for 12 consecutive weeks.

Exclusion Criteria:

* Pregnant women
* Participants who had undergone spinal surgery
* Participants who complained of neurological symptoms, such as parasthesia in lower limbs
* Participants who suffered from severe controlled hypertension
* Participants who were involved in other exercise, such as Pilates
* Participants who were not willing/unable to commit to attending the Pilates sessions for the duration of study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Questionnaire 1 | To be distributed to patients prior to an intervention.
  The perception of Pilates as a treatment in the management of Low Back Pain.
Questionnaire 2 | To be given immediately after completing the intervention programme.
  Post Pilates programme feedback questionnaire.

SECONDARY OUTCOMES:
Numerical Pain Rating Scale | Up to 1 year since start of the intervention.
  It is a self-reported measure where individuals are asked to rate their pain on a numerical scale. Zero means 'no pain' and 10 means 'the worst possible pain'.
Quebec Back Pain Disability Scale | Up to 1 year since start of the intervention.
  It is a tool designed to assess the impact of chronic pain on daily functioning and activities, particularly focusing on disability associated with pain conditions. The score disability level range from: 0 - 4 No disability, 5 - 14 Mild disability, 15 - 24 Moderate disability, 25 - 34 Severe disability and 35 - 50 Completely disabled.
RAND 36-Item Health Survey | Up to 1 year since start of the intervention.
  It is a widely used health survey measuring various aspects of physical and mental well-being to assess an individual's health-related quality of life. Possible scores range from 0 to 100, with higher scores representing better health status.
Hospital Anxiety and Depression Scale | Up to 1 year since start of the intervention.
  It is a self-assessment tool used to measure anxiety and depression levels in patients within a medical care setting. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level.

CONTACTS AND LOCATIONS:
Overall Officials: Mr Tonio Agius, Principal Investigator — Principal Supervisor; Anabel Sciriha, Principal Investigator — Co-supervisor

IPD SHARING:
Plan to Share IPD: No